CLINICAL TRIAL: NCT05624944
Title: An Open-label Pharmacokinetic Study of TS-142 in Patients with Hepatic Impairment
Brief Title: A Pharmacokinetic Study of TS-142 in Patients with Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS142-303
Record Dates: First submitted 2022-11-11; First posted 2022-11-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-12

CONDITIONS: Patients with Mild or Moderate Hepatic Impairment
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mild hepatic impairment (Experimental): Patients with mild hepatic impairment will receive a single-dose of 5 mg of TS-142
  Interventions: Drug: TS-142 5 mg
- Moderate hepatic impairment (Experimental): Patients with moderate hepatic impairment will receive a single-dose of 5 mg of TS-142
  Interventions: Drug: TS-142 5 mg
- Normal hepatic function (Experimental): Subjects with normal hepatic function will receive a single-dose of 5 mg of TS-142
  Interventions: Drug: TS-142 5 mg

INTERVENTIONS:
Drug: TS-142 5 mg — Single-dose of 5 mg of TS-142

SUMMARY:
This is an open-label pharmacokinetic study of TS-142 in patients with hepatic impairment

ELIGIBILITY:
Inclusion Criteria:

<Inclusion criteria for patients with hepatic impairment>

1. Japanese male and female who are aged 18 to 75 years at the time of informed consent
2. Patients with cirrhosis or chronic hepatic impairment
3. Patients classified as Child-Pugh classification A (mild) or B (moderate) by the principal investigator or sub-investigator at the screening test Other protocol defined inclusion criteria could apply.

<Inclusion criteria for subject with normal hepatic function>

1. Japanese male and female who are aged 18 to 75 years at the time of informed consent
2. Body Mass Index (BMI) between 18.5 and 35.0 at the screening test Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

<Exclusion criteria for patients with hepatic impairment>

1. Patients who have a history of liver resection or liver transplant
2. Patients with hepatic encephalopathy of grade II or higher
3. Patients with epidermal growth factor receptor (eGFR) less than 45 mL/min/1.73 m2 at the screening test Other protocol defined exclusion criteria could apply.

<Exclusion criteria for subjects with normal hepatic function>

1. Subjects who are judged to have any disease by the principal investigator or sub-investigator
2. Subjects with eGFR less than 60 mL/min/1.73 m2 at the screening test Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | Predose and up to 48 hours postdose
  Plasma concentration of unchanged form and its metabolite
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Maximum plasma concentration of unchanged form and its metabolite (Cmax)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Time to maximum plasma concentration of unchanged form and its metabolite (tmax)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Area under the plasma concentration-time curve extrapolated to infinity of unchanged form and its metabolite (AUCinf)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of unchanged form and its metabolite (AUC0-last)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Terminal elimination rate constant of unchanged form and its metabolite (λz)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Elimination half-life of unchanged form and its metabolite (t1/2)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Apparent volume of distribution based on the terminal phase of unchanged form (Vz/F)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Apparent total body clearance of unchanged form (CL/F)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Plasma unbound fraction of unchanged form and its metabolite (fu)
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Maximum plasma concentration adjusted by unbound fraction of unchanged form (Cmax(unbound))
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Area under the plasma concentration-time curve extrapolated to infinity adjusted by unbound fraction of unchanged form (AUC(unbound))
Pharmacokinetic parameters | Predose and up to 48 hours postdose
  Apparent total body clearance adjusted by unbound fraction of unchanged form (CL(unbound)/F)

SECONDARY OUTCOMES:
Incidence of adverse events | From administration of investigational product through 10 days after administration of investigational product
  "Adverse event" refers to any unfavorable or unintended disease or symptom thereof (including abnormal laboratory tests values) occurring in a subject who has been administered an investigational product, whether or not there is a causal relationship with the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No